CLINICAL TRIAL: NCT01528085
Title: An Open Label Phase II Study to Evaluate the Efficacy and Safety of Induction and Consolidation Therapy With Nilotinib in Combination With Chemotherapy in Patients Aged 55 Years and Over With Philadelphia Chromosome Positive (Ph+ or BCR-ABL+) Acute Lymphoblastic Leukemia (ALL)
Brief Title: Evaluation of Efficacy and Safety of Nilotinib in Combination With Chemotherapy in Elderly Patients With Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Heike Pfeifer MD, Dr.med., Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EWALL-PH-02; 2010-022855-46 (EudraCT Number)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Philadelphia Chromsome Positive Acute Lymphoblastic Leukemia
Keywords: Philadelphia chromsome; BCR-ABL; ALL; acute lymphoblastic leukemia; Nilotinib; Tasigna
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nilotinib — Nilotinib, p.o Chemotherapy (Dexamethasone, Methotroxate, Cyclophosphamide (optional), Vincristine, Vindesine, Cytarabine, 6-Mercapto-Purine)
  Other Names: Tasigna

SUMMARY:
The goal of this trial is to evaluate the efficacy and the tolerance of the combination of nilotinib with chemotherapy in the front-line setting as induction and consolidation therapy in Ph+ ALL patient aged 55 years and over. A European consensus has been reached to adopt a common chemotherapeutic schedule for patients aged 55 years and over. This schedule will be used in this trial with the addition of nilotinib as concomitant therapy during induction, consolidation and maintenance. The patients will be prospectively monitored for minimal residual disease and bcr-abl tyrosine kinase domain mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 55 years
2. Philadelphia chromosome- or BCR-ABL positive acute lymphoblastic leukemia
3. Not previously treated except with corticosteroids or single dose vincristine (three doses cyclophosphamide accepted)
4. With or without documented CNS involvement
5. WHO performance status < 2
6. Normal serum levels > LLN (lower limit of normal) of potassium, magnesium, total calcium corrected for serum albumin; or corrected to within normal limits with supplements, prior to the first dose of study medication
7. Signed written inform consent
8. Molecular evaluation for BCR-ABL performed
9. Willingness of male subjects whose sexual partners are women of child-bearing potential (WOCBP), to use an effective form of contraception (pearl index < 1%), such as complete sexual abstinence, combined oral contraceptive, hormone IUCD, vaginal hormone ring, transdermal contraceptive patch, contraceptive implant or depot contraceptive injection in combination with a second method of contraception like a condom or a cervical cap / diaphragm with spermicide or surgical sterilisation (vasectomy) in male patients during the study and at least 6 months thereafter. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or surgical sterilization or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Patient previously treated with tyrosine kinase inhibitors
2. Known impaired cardiac function, including any of the following:

   * LVEF < 45%
   * Complete left bundle branch block
   * Right bundle branch block plus left anterior hemiblock, bifascicular block
   * Use of a ventricular-paced pacemaker
   * Congenital long QT syndrome
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (< 50 beats per minute)
   * QTcF>450 msec on screening ECG. If QTc > 450 msec and electrolytes are not within normal ranges before nilotinib dosing, electrolytes should be corrected and then the patient rescreened for QTcF criterion.
   * Myocardial infarction with 12 months prior to starting nilotinib
   * Other clinical significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)
3. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
4. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory) or known infection with Hepatitis B or C
5. Treatment with any, other investigational agent or participating in another trial within 30 days prior to entering this study
6. Inadequate hepatic functions defined as ASAT or ALAT > 2,5 times the institutional upper limit of normal or > 5 times ULN if considered due to leukemia
7. Total bilirubin > 2 fold the institutional upper limit unless considered to be due to organ involvement by the leukemia or to M. Gilbert / M. Meulengracht
8. Concurrent severe diseases which exclude the administration of therapy
9. Past history of acute or chronic pancreatits
10. Patients unwilling or unable to comply with the protocol.e branch block; Right bundle branch block plus left anterior hemiblock, bifascicular block; Use of a ventricular-paced pacemaker; congenital long QT syndrome

    * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
    * Clinically significant resting bradycardia (< 50 beats per minute)
    * QTcF>450 msec on screening ECG. If QTc > 450 msec and electrolytes are not within normal ranges before nilotinib dosing, electrolytes should be corrected and then the patient rescreened for QTcF criterion.
    * Myocardial infarction with 12 months prior to starting nilotinib
    * Other clinical significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)

      * Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
      * Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory) or known infection with Hepatitis B or C
      * Treatment with any, other investigational agent or participating in another trial within 30 days prior to entering this study
      * Inadequate hepatic functions defined as ASAT or ALAT > 2,5 times the institutional upper limit of normal or > 5 times ULN if considered due to leukemia
      * Total bilirubin > 2 fold the institutional upper limit unless considered to be due to organ involvement by the leukemia or to M. Gilbert / M. Meulengracht
      * Concurrent severe diseases which exclude the administration of therapy
      * Past history of acute or chronic pancreatits
      * Patients unwilling or unable to comply with the protocol.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-01; Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of a nilotinib-based induction and consolidation therapy | after 12 months
  rate of patients without event

SECONDARY OUTCOMES:
complete haematological remission | after induction treatment (week 5)
  The rate of complete haematological remission after induction treatment
major molecular response in bone marrow
  major molecular response defined by a BCR-ABL/ABL < 0.1% in bone marrow
complete molecular response
  complete molecular response defined by a BCR-ABL/ABL < 0.001% in bone marrow
undetectable BCR-ABL level
  The proportion of patients with confirmed undetectable BCR-ABL level with a test sensitivity of at least 4.5 log.
Event free survival
Relapse free survival
Progression free survival
T315I or p-loop Mutations
  Detection of a T315I or p-loop BCR-ABL TK domain mutation
molecular relapse or progression
  The proportion of patients with molecular relapse or progression
Overall survival
Tolerability
  Tolerability as determined by descriptive assessment of adverse events and discontinuation due to treatment-related SAEs
Death during induction | End of induction (week 5)
  (all patients who started treatment)
Death in complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Heike Pfeifer, Dr.med., Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (69):
- France (41):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - CHU d'Amiens - Hôpital Sud, Amiens
  - Chu Angers, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Brest - Hôpital Morvan, Brest
  - "CHU Cote de nacre ", Caen
  - CHU Estaing, Clermont-Ferrand
  - AP-HP - Hôpital Henri Mondor, Créteil
  - CHRU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CH de Versailles - Hôpital André Mignot, Le Chesnay
  - Groupe Hospitalier de l'Institut Catholique de Lille, hôpital Saint-Vincent, Lille
  - CHRU de Lille, Lille
  - C H U de Limoges - Hôpital Dupuytren, Limoges
  - Institut Paoli-Calmettes, Marseille
  - CH de Meaux, Meaux
  - Hôpital Saint-Eloi, Montpellier
  - CH de Mulhouse - Hôpital Emile Muller, Mulhouse
  - CHU Hôtel Dieu, Nantes, Nantes
  - CHU de Nice - Hôpital l'Archet 1, Nice
  - CHR d'Orléans - Hôpital La Source, Orléans
  - AP-HP - Hôpital Saint Louis, Paris
  - AP-HP - Hôpital SAINT-ANTOINE, Paris
  - AP-HP - Hôpital Necker, Paris
  - CH de Perpignan - Hôpital Saint-Jean, Perpignan
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital La Milétrie, Poitiers
  - CH de la Région d'Annecy, Pringy
  - CHU de Reims - Hôpital Robert Debré, Reims
  - CHU de Rennes, Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen, Rouen
  - CHU de La Réunion - Hôpital Félix Guyon, Saint-Denis
  - CHRU de Strasbourg - Hôpital Hautepierre, Strasbourg
  - HIA Sainte Anne, Toulon
  - "Institut Universitaire du Cancer (CHU de Toulouse - Hôpital Purpan)", Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours
  - Centre Hospitalier de Valenciennes, Valenciennes
  - CHU de Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
- Germany (22):
  - Robert Bosch Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Klinikum der Universität Regensburg, Regensburg, Bavaria
  - University Hospital of Frankfurt, Medical Dept. II, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinik Münster, Münster, North Rhine-Westphalia
  - Universitätsklinik Dresden, Dresden, Saxony
  - Uniklinik Aachen, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Göttingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universität Leipzig, José-Carreras-Haus, Leipzig
  - Universitätskliniken Mainz, Mainz
  - Klinikum Mannheim, Mannheim
  - Universitätsklinikum Großhadern, München
  - Klinikum Nürnberg Nord, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Universität Rostock, Rostock
  - Medizinische Universitätsklinik Ulm, Ulm
  - Universität Würzburg, Würzburg
- Spain (6):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Germans Trias i Pujol (ICO - Badalona), Barcelona
  - Hospital Universitario 12 de Octubre (Madrid), Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío (Sevilla), Seville
  - Hospital Universitario y Politécnico La Fe (Valencia), Valencia

REFERENCES:
- See also: Trial register of University Cancer Center Frankfurt, additional trial information — https://www.uct-frankfurt.de/fuer-aerzte/klinische-studien.html